CLINICAL TRIAL: NCT06803992
Title: Induction of Labor in Women With Unfavorable Cervix at Term - Comparison of Propess Versus Prostaglandin E2 Vaginal Gel and Extra-amniotic Balloon Catheter
Brief Title: Induction of Labor - Comparison Propess With Prostaglandin E2 Vaginal Gel and Balloon Catheter
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Zohar Nachum, professor, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 79-23
Record Dates: First submitted 2025-01-19; First posted 2025-01-31 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-01

CONDITIONS: Induction of Labor

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propess pessary (Experimental): Placement of a slow-release 10 mg dinoprostone insert (propess) in the posterior fornix for up to 24 hours until labor initiation or favorable cervix, followed by amniotomy and oxytocin administration. In a case of failure, induction of labor will be done with either PGE2 gel and/or Foley catheter.
  Interventions: Drug: Dinoprostone vaginal insert
- Sequential PGE2 vaginal gel and Foley catheter balloon (Experimental): Insertion of 1 mg dinoprostone (PGE2) vaginal gel to the posterior fornix with reassessment up to 6 hours later. If the Bishop score is still less than 5 and there are no more than 4 contractions in 20 minutes of monitoring, an additional PGE2 vaginal gel of 2 mg is inserted. If there are more than 4 contractions in 20 minutes of monitoring or if after up to 6 hours there will be low Bishop score, a 60 ml Foley catheter balloon is placed for 6 to 12 hours or until spontaneous expulsion. When the cervix is favorable, amniotomy and oxytocin administration are followed.
  In a case of a failure, induction of labor with Propess will be conducted.
  Interventions: Combination Product: Dinoprostone gel and Foley catheter balloon

INTERVENTIONS:
Drug: Dinoprostone vaginal insert — Described in the arm descriptions
  Other Names: Propess
  Arms: Propess pessary
Combination Product: Dinoprostone gel and Foley catheter balloon — Described in the arm descriptions
  Arms: Sequential PGE2 vaginal gel and Foley catheter balloon

SUMMARY:
One of every four births in the Western world is induced, usually due to the risk of maternal and fetal morbidity. There are several methods of labor induction, pharmacological and mechanical. In cases of unfavorable cervix (Bishop score is below 5), cervical ripening can be induced by either prostaglandins E2 (slow release 10 mg dinoprostone insert (propess) or vaginal gel 1-2 mg) or mechanically by Foley catheter balloon (FCB).

The efficacy of labor induction of propess versus vaginal gel combined with FCB was not studied previously.

The goal of this randomized controlled trial is to compare the efficacy of propess versus PGE2 vaginal gel combined with FCB in women with singletons undergoing labor induction at term. The main question it aims to answer is to compare the time from the beginning of labor induction until delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at term (37 weeks of gestation or more) with singleton
* pregnancies that are intended for IOL.
* Initial bishop score <5
* No contraindications to receive either treatment.
* Women who will give informed consent to be included in the study.
* Women at or over the age of 18.

Exclusion Criteria:

* Women with a known hypersensitivity or contraindications to Propess / PGE2.
* Parity 5 or more
* Labor contractions more than 4 in 20 min
* Glaucoma
* History of previous uterine surgery
* Hypersensitivity to prostaglandins
* Vaginal delivery is contraindicated
* Active cardiac, renal, pulmonary, or hepatic disease
* Severe asthma or pulmonary disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
comparing the duration of induction-to-vaginal delivery | from enrollment until final outcome - a month
  measuring the duration of Induction-of-labor by Propess versus the combined use of PGE2 gel and balloon catheter by induction-to-vaginal delivery interval from the beginning of the induction according to the chosen patient protocol and until vaginal delivery.

SECONDARY OUTCOMES:
rate of vaginal delivery in 24 and 48 hours from IOL | from enrollment until final outcome - a month
  the number of participants who had vaginal delivery in 24 and 48 hours from the beginning of the induction-of-labor for both protocols
Number of Participants with Treatment-Related Adverse Events | from enrollment until final outcome - a month
  Maternal -gathering the numbers of participants who had adverse events such as chorioamnionitis, endometritis, postpartum hemorrhage, uterine rupture, Neonatal -gathering the numbers of participants who had adverse events such as uterine hypertonia (contractions exceeding more than two minutes in duration) and/or tachysystole (more than 5 contractions in 10 minutes, averaged over a 30-minute period) with and without decelerations, non-reassuring fetal heart rate according to fetal monitoring, meconium-stained amniotic liquor, umbilical artery pH less than 7.1, Apgar score less than 7 at 5 min, postpartum transfer to neonatal intensive care unit, infection of the newborn
rate of Induction success | from enrollment until final outcome - a month
  the number of participants who had ceasarean section
rate o Cervical ripening success | from enrollment until final outcome - a month
  the duration from the beginning of the induction to bishop score 5

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Nachum, Professor, Study Director — Emek Medical Center
Locations (1):
- Emek medical center, Afula, Israel